CLINICAL TRIAL: NCT05283122
Title: Mostafa Maged Technique to Control and Prevent the Post-Partum Bleeding From the Lower Uterine Segment in Placenta Previa Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mostafa Maged Ali, Principal investigator, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R 207
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Placenta Previa
Keywords: Mostafa Maged technique; placenta previa; lower uterine segment; caeserian section
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: primigravida pregnant patients with placenta previa conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Mostafa Maged technique to prevent and control post-partum bleeding in placenta previa cases (Experimental): primigravida patients with placenta previa conditions and their ages between ( 18 - 30 ) years old
  Interventions: Procedure: Mostafa Maged Technique

INTERVENTIONS:
Procedure: Mostafa Maged Technique — pfannestiel incision . dissection of the bladder downwards , and Ligation of the uterine arteries on both sides then , we turn over the upper part of the lower uterine segment onto the lower part of the lower uterine segment from the inside of uterine cavity .We do this turnover (flipping ) by our hands and holding the imaginary line by two Allis forceps and by making three knots by three needles in the lower edge of the uterine incision and we enter the needles of simultaneously into the lower segment through the uterine cavity , at the same level of , the inside wall of lower uterine segment to drag the upper (half) part of the lower uterine segment on the lower part of lower uterine segment ( sandwich - like ) Third , we stitch the both sides of the flipped lower uterine segment , then we do plication of the anterior lower uterine segments to strengthen the wall of the flipped lower uterine segment and place a drain in the doglus pouch

SUMMARY:
Post - partum haemorrhage is still a headache to all obstetricians around the whole world . Every obstetrician exerts his own full effort to control bleeding which can occur post-partum by applying all maneuvers to preserve the fertility and the uterus for the patient .

demonstration of ( Mostafa Maged ) technique is applied to control and prevent post-partum haemorrhage . It is so simple maneuver and easy to be applied within short period of time .Satisfactory hemostasis can be assessed after application .

DETAILED DESCRIPTION:
1. pfannestiel incision .
2. dissection of the bladder downwards , and then making an incision in the lower segment of the uterus , then the uterus is evacuated from the fetus and placenta .
3. Ligation of the uterine arteries on both sides is applied before proceeding and after the extraction of fetus and placenta .

5) The lower segment was bleeding so trying to do bimanual compression of the anterior and posterior parts of lower uterine segments to test if Mostafa Maged technique is useful in these cases or not (( by observing if the bleeding is minimized or stopped or not by compression )) as if it is minimized so our technique has a high chance to be effective .

6) The whole technique depends on the anterior lower uterine segment by dividing the anterior lower uterine segment by an imaginary line in two halves , then , turning over (flipping ) the upper part of the lower uterine segment onto the lower part of the lower uterine segment from the inside of uterine cavity .

7) doing this turnover (flipping ) by the hands and holding the imaginary line by two Allis forceps and by making three knots by three needles in the lower edge of the uterine incision and entering the needles of (absorbable 70 mm rounded-bodied vicryl 1 ) simultaneously into the lower segment through the uterine cavity , at the same level of , the inside wall of lower uterine segment in order to drag the upper (half) part of the lower uterine segment on the lower part of lower uterine segment ( sandwich - like ) , and after this maneuver the bleeding is re-evaluated again .

8) Third , stitching the both sides of the flipped lower uterine segment by ( absorbable 70 mm rounded-bodied vicryl 1 ) , then doing plication of the anterior lower uterine segments to strengthen the wall of the flipped lower uterine segment and secure the tension .

9) Fourth , closing the caeserian scar by suturing the already-flipped lower uterine segment onto the upper uterine segment .

10) placing a drain in the doglus pouch

ELIGIBILITY:
Inclusion Criteria:

* pregnant primigravida patients with placenta previa
* 18 to 30 years old

Exclusion Criteria:

* patients with bleeding disorders
* smokers
* morbid obese patients

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
primary post-partum bleeding | twenty-four hours post-partum
  prevention and management of bleeding from lower segment ....estimation of number of pads used during section to estimate blood loss ... and to assess the number of blood loss postpartum roughly visually

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum general hospital and Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No